CLINICAL TRIAL: NCT03106272
Title: Anti-Mullerian Hormone Dynamics During Natural Cycle Using Automated Assay
Brief Title: Evaluating the AMH Levels During Natural Cycle
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Medical Director, ART Fertility Clinics LLC
Other Study IDs: 1611-ABU-083-HF
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-07

CONDITIONS: Anti-Mullerian Hormone Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anonymized samples will be obtained, nurses are those charged with patient blood extraction by venipuncture from a vein in the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe AMH serum levels dynamics during natural cycle using an automated assay.

DETAILED DESCRIPTION:
The potential benefit would be using an automated assay for AMH, the dynamics of serum levels during the natural cycle and to check the inter-cycle variations.

Because of the many clinical decisions that are based on AMH levels alone the results of this study could bring reassurance to the continuous use of AMH in daily practice. More importantly, no studies to date have been performed on the newer automated assays evaluating variability of AMH levels.

ELIGIBILITY:
Inclusion Criteria:

* Women with written informed consent.
* Women between ≥ 18 and ≤ 37 years of age.
* BMI between 18 and 28.
* Normal physical examination and pelvic exam.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* History of any disease/iatrogenic intervention which could have had an impact on the ovarian reserve (e.g. ovarian surgery, chemotherapy, radiation of the pelvis, endometriosis)
* Intake of OCP for the two last menstrual cycles.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women.
Study Population: Healthy women with regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
AMH serum levels dynamic | 9months
  In order to describe each hormone and its dynamics, will determine mean and standard deviations in each time and it will be represented with boxplot figures.
  Moreover,the investigator will define polynomial interpolation for dynamic values and each hormone will be represented with mean polynomial interpolation and variance band

SECONDARY OUTCOMES:
Inter-cycle AMH variations | 9months
  inter-cycle variability of AMH across two cycles is concluded independently that AMH varies a little between cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Human Fatemi, Medical D., Principal Investigator — IVI Middle East Fertility Clinic LLC
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Anderson RA, Anckaert E, Bosch E, Dewailly D, Dunlop CE, Fehr D, Nardo L, Smitz J, Tremellen K, Denk B, Geistanger A, Hund M. Prospective study into the value of the automated Elecsys antimullerian hormone assay for the assessment of the ovarian growing follicle pool. Fertil Steril. 2015 Apr;103(4):1074-1080.e4. doi: 10.1016/j.fertnstert.2015.01.004. Epub 2015 Feb 11. PMID 25681853
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Background] Hehenkamp WJ, Looman CW, Themmen AP, de Jong FH, Te Velde ER, Broekmans FJ. Anti-Mullerian hormone levels in the spontaneous menstrual cycle do not show substantial fluctuation. J Clin Endocrinol Metab. 2006 Oct;91(10):4057-63. doi: 10.1210/jc.2006-0331. Epub 2006 Jun 27. PMID 16804046
- [Background] La Marca A, Grisendi V, Griesinger G. How Much Does AMH Really Vary in Normal Women? Int J Endocrinol. 2013;2013:959487. doi: 10.1155/2013/959487. Epub 2013 Nov 19. PMID 24348558
- [Background] La Marca A, Stabile G, Artenisio AC, Volpe A. Serum anti-Mullerian hormone throughout the human menstrual cycle. Hum Reprod. 2006 Dec;21(12):3103-7. doi: 10.1093/humrep/del291. Epub 2006 Aug 21. PMID 16923748
- [Background] Lambert-Messerlian G, Plante B, Eklund EE, Raker C, Moore RG. Levels of antimullerian hormone in serum during the normal menstrual cycle. Fertil Steril. 2016 Jan;105(1):208-13.e1. doi: 10.1016/j.fertnstert.2015.09.033. Epub 2015 Oct 23. PMID 26477497
- [Background] Overbeek A, Broekmans FJ, Hehenkamp WJ, Wijdeveld ME, van Disseldorp J, van Dulmen-den Broeder E, Lambalk CB. Intra-cycle fluctuations of anti-Mullerian hormone in normal women with a regular cycle: a re-analysis. Reprod Biomed Online. 2012 Jun;24(6):664-9. doi: 10.1016/j.rbmo.2012.02.023. Epub 2012 Mar 9. PMID 22503280
- [Background] Rustamov O, Smith A, Roberts SA, Yates AP, Fitzgerald C, Krishnan M, Nardo LG, Pemberton PW. The measurement of anti-Mullerian hormone: a critical appraisal. J Clin Endocrinol Metab. 2014 Mar;99(3):723-32. doi: 10.1210/jc.2013-3476. Epub 2013 Jan 1. PMID 24423305
- [Background] Seifer DB, Maclaughlin DT. Mullerian Inhibiting Substance is an ovarian growth factor of emerging clinical significance. Fertil Steril. 2007 Sep;88(3):539-46. doi: 10.1016/j.fertnstert.2007.02.014. Epub 2007 Jun 7. PMID 17559842
- [Background] Sowers M, McConnell D, Gast K, Zheng H, Nan B, McCarthy JD, Randolph JF. Anti-Mullerian hormone and inhibin B variability during normal menstrual cycles. Fertil Steril. 2010 Sep;94(4):1482-1486. doi: 10.1016/j.fertnstert.2009.07.1674. Epub 2009 Dec 6. PMID 19969291
- [Background] Streuli I, Fraisse T, Pillet C, Ibecheole V, Bischof P, de Ziegler D. Serum antimullerian hormone levels remain stable throughout the menstrual cycle and after oral or vaginal administration of synthetic sex steroids. Fertil Steril. 2008 Aug;90(2):395-400. doi: 10.1016/j.fertnstert.2007.06.023. Epub 2007 Oct 24. PMID 17919608
- [Background] Tsepelidis S, Devreker F, Demeestere I, Flahaut A, Gervy Ch, Englert Y. Stable serum levels of anti-Mullerian hormone during the menstrual cycle: a prospective study in normo-ovulatory women. Hum Reprod. 2007 Jul;22(7):1837-40. doi: 10.1093/humrep/dem101. Epub 2007 May 7. PMID 17485437
- [Background] van Disseldorp J, Lambalk CB, Kwee J, Looman CW, Eijkemans MJ, Fauser BC, Broekmans FJ. Comparison of inter- and intra-cycle variability of anti-Mullerian hormone and antral follicle counts. Hum Reprod. 2010 Jan;25(1):221-7. doi: 10.1093/humrep/dep366. Epub 2009 Oct 19. PMID 19840990
- [Background] van Rooij IA, Bancsi LF, Broekmans FJ, Looman CW, Habbema JD, te Velde ER. Women older than 40 years of age and those with elevated follicle-stimulating hormone levels differ in poor response rate and embryo quality in in vitro fertilization. Fertil Steril. 2003 Mar;79(3):482-8. doi: 10.1016/s0015-0282(02)04839-2. PMID 12620425